CLINICAL TRIAL: NCT04932447
Title: Time-efficient Inspiratory Muscle Strength Training for Improving Blood Pressure and Vascular Function in Older Adults With Sleep Disordered Breathing
Brief Title: Breathing Training for Improving Cardiovascular Health in Older Adults With Sleep Apnea
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH); University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Elizabeth Fiona Bailey, PhD, Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1200000220; 1R01AG065346-01A1 (NIH)
Record Dates: First submitted 2021-04-27; First posted 2021-06-21 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea; Hypertension
Keywords: Inspiratory Muscle Strength Training; Blood Pressure; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated using a 1:1 ratio to A) High-Intensity Training Group (75 % maximal inspiratory pressure) or B)Low-Intensity Training Group (15% maximal inspiratory pressure)
Who Masked: Participant, Investigator
Masking Description: This is a randomized double-blinded clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training Group A (Experimental): Participants will perform their respiratory training (high-intensity, low-volume IMST) on a hand-held respiratory training device.
  Interventions: Behavioral: Inspiratory Muscle Strength Training
- Training Group B (Sham Comparator): Participants will perform their respiratory training (low-intensity, low-volume IMST) on a hand-held respiratory training device.
  Interventions: Behavioral: Inspiratory Muscle Strength Training

INTERVENTIONS:
Behavioral: Inspiratory Muscle Strength Training — 30 breaths/ day, 5 days/week for 24 weeks.

SUMMARY:
This clinical research study will investigate the effects of respiratory strength training on blood pressure and cardiovascular health in adults who are 50 years of age and older and have been diagnosed with moderate or severe obstructive sleep apnea.

DETAILED DESCRIPTION:
Exercise has well-documented benefits for systolic blood pressure (SBP) and cardiovascular health. Whereas current guidelines advocate ~150 min moderate intensity exercise/week, our preliminary data show ~5 min/day of inspiratory muscle strength training (IMST) for 6 weeks lowers casual (resting) SBP by ~12 mmHg.

This simple approach to lowering BP could be applied to almost any population however we are studying IMST in older adults with obstructive sleep apnea (OSA). OSA is an ideal population to target because OSA prevalence is growing and because snoring and apneas result in chronic intermittent hypoxemia that drives sympathetic nervous system (SNS) hyperactivity, endothelial dysfunction and hypertension. These substantive risks for cardiovascular disease are compounded by poor adherence to the mainstay treatment continuous positive airway pressure (<50%), obesity, fatigue and a robust intolerance for exercise.

Our findings in healthy young adults (n=50) show IMST-related reductions in BP are mediated by decreases in systemic vascular resistance, suggesting changes in vascular tone and function. Consistent with this hypothesis, our results from a pilot clinical trial in adults with OSA (n=24) show IMST-related reductions in plasma norepinephrine levels (PNE) and muscle sympathetic nerve activity (MSNA), both markers of SNS activity. Our preliminary mechanistic assessments indicate IMST may lower circulating concentrations of other vasoconstrictor factors and increase nitric oxide (NO)-mediated endothelium-dependent dilation. And, findings in a novel endothelial cell culture model, point to increases in NO and declines in reactive oxygen species (ROS) and oxidative stress. However, it is unknown if: 1) IMST lowers casual and 24-h (ambulatory) SBP in older adults with OSA; 2) the reductions in SBP are long-lasting; 3) arterial stiffness, NO-mediated endothelial dilation and/or oxidative stress are improved; and 4) if adherence in this population is high long term.

In this randomized, double-blind clinical trial we will establish the efficacy of high-intensity IMST (75% maximum inspiratory pressure, [PImax]) 5 days/week for 24 weeks vs. low-intensity IMST (15%PImax) (n=61/group) for lowering SBP in adults (>50 years) with above normal BP and OSA. We hypothesize that IMST will lower SBP via reductions in SNS activity and circulating vasoconstrictor factors, improvements in vascular function, and reductions in oxidative stress/inflammation and that reductions in SBP will be sustained 4 and 12 weeks post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 and older
* Ability to understand study procedures and to comply with them for the entire length of the study
* Ability to provide informed consent;
* Willing to accept random assignment to condition
* AHI ≥15
* Individuals with who are unwilling or unable to adhere to CPAP
* Individuals who are adherent to CPAP therapy (i.e., 4 hours/night on 70%/nights over 30 days in the first 3 months of initial usage)
* Individuals who are adherent to mandibular advancement device each night
* Above-normal SBP (i.e., SBP ≥120)
* BMI ≤40 kg/m2
* Weight stable in the prior 3 months (<3.0 kg weight change) and willing to remain weight stable throughout the study
* No change in anti-hypertensive medications or other medications (prescription or dosing) in the prior 3 months and willingness to maintain current medication regimen throughout the study
* Absence of unstable clinical disease as determined by medical history, physical examination, and blood chemistries
* Total cholesterol <240 mg/dL
* Fasting plasma glucose <300 mg/dL

Exclusion Criteria:

* Age <50
* AHI <15
* Individuals with central or mixed sleep disordered breathing
* Severe hypoxemia (<80% for >10% of recording time) during sleep
* ESS >15
* SBP ≥160 or DBP ≥120
* Current smoker
* Chronic overt and poorly controlled medical condition (e.g., diabetes, chronic kidney disease, cancer, congestive heart failure)
* Cheyne-Stokes Respiration
* Alcohol or illegal drug dependence or abuse
* Uncontrolled thyroid disease or change in thyroid medication within previous 3 months
* Regular/vigorous aerobic exercise (> 4 bouts/week, >30 min/bout at high workload >6 METS)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline casual Systolic Blood Pressure at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  The primary endpoint is casual (resting) systolic blood pressure (SBP) measured by both relative and absolute changes from baseline. SBP will be assessed in accordance with American College of Cardiology/American Heart Association guidelines. Measurements will be taken using an automated oscillometric sphygmomanometer and will be performed in triplicate over the brachial artery of the non-dominant arm after 5 minutes of quiet rest, with 1 minute of recovery between measures. SBP will be defined as the average of the 3 pressures.

SECONDARY OUTCOMES:
Change from baseline 24-hour Ambulatory Systolic Blood Pressure at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  The secondary endpoint is 24-hour ambulatory systolic blood pressure measured by both relative and absolute changes from baseline. We will obtain continuous measures of systolic and diastolic blood pressure over a 24-h period with an FDA approved and European Society of Hypertension validated Non-Invasive Ambulatory Blood Pressure monitor. Blood pressure data will be broken into daytime (16 hour) and nighttime (8 hour) segments according to participants' individual sleep-wake cycles. Mean systolic and diastolic blood pressures (mmHg) will be calculated for the daytime and nighttime periods to evaluate circadian systolic and diastolic blood pressure profiles.
Change from baseline Plasma Norepinephrine at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  The secondary endpoint is Plasma Norepinephrine (PNE), a marker of sympathetic activity, measured by both relative and absolute changes from baseline. PNE will be determined from venous (antecubital area) blood samples and quantified via high performance liquid chromatography (HPLC). PNE will be measured following a fasting blood draw collected between the hours of 7:00 and 10:00 am, preceded by 30 minutes supine rest in a quiet, temperature-controlled room.

OTHER OUTCOMES:
Change from baseline Nitric Oxide-mediated Endothelial Dependent Dilation (EDD) and suppression of EDD by oxidative stress at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  Brachial artery Flow Mediated Dilation (BA-FMD), a well-established measure of NO-mediated endothelial function, will be measured by both relative and absolute changes from baseline. BA-FMD will be determined using high-resolution ultrasonography and analyzed with a commercially available software package. An ultrasound probe will be placed 3-6 cm proximal to the antecubital crease on the right arm and a baseline image of the right brachial artery will be obtained. Following baseline, reactive hyperemia will be produced by inflating a rapid-inflating blood pressure cuff. Brachial artery diameter change will be measured for 2 minutes following 5-min of forearm blood flow occlusion. To determine tonic oxidative stress-mediated suppression of BA-FMD the difference in BA-FMD observed with and without supraphysiological infusion of vitamin C will be measured.
Change from baseline Carotid-Femoral Pulse Wave Velocity at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  Carotid-Femoral Pulse Wave Velocity (CFPWV) will be will be measured by both relative and absolute changes from baseline. CFPWV determined via transcutaneous tonometry of the carotid and femoral arteries will be recorded consecutively. The transit time (TT) between the foot and the pressure waves measured at each location will be determined by using the R-wave of the ECG recording taken during the tonometry procedure as a timing reference.
Change from baseline vasoconstrictor factors at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  Circulating levels of vasoconstrictor molecules ET-1 and Ang-2 will be measured by both relative and absolute changes from baseline. ET-1 and Ang-2 will be assessed by enzyme-linked immunosorbent assays (ELISA.)
Change from baseline influence of circulating factors on endothelial Nitric Oxide and Reactive Oxygen Species at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  We asses the influence of circulating factors on endothelial NO and ROS by measuring both relative and absolute changes from baseline. We will expose cultured human umbilical vein endothelial cells (HUVECs, American Type Culture Collection) ex vivo, to media conditioned with serum drawn from participants' blood samples to determine if IMST improves endothelial function via changes in circulating factors that increase endothelial cell NO production and/or reduce endothelial ROS production.
Change from Baseline Muscle Sympathetic Nerve Activity at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  Muscle Sympathetic Nerve Activity (MSNA) will be measured by both relative and absolute changes from baseline. MSNA recorded via microelectrode inserted into the common peroneal nerve immediately posterior to the fibular head. Electrode placement will be confirmed via electrical stimulation. Burst frequency (burst/min) and burst incidence (bursts per 100 heart beats) and total activity (mean burst area /min) will be obtained from the integrated MSNA signal.
Change from Baseline Casual Diastolic Blood Pressure (DBP) at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  Casual (resting) measures of diastolic blood pressure will be assessed in accordance with American College of Cardiology/American Heart Association guidelines. Measurements will be taken using an automated oscillometric sphygmomanometer and will be performed in triplicate over the brachial artery of the non-dominant arm after 5 minutes of quiet rest, with 1 minute of recovery between measures. DBP will be defined as the average of the 3 pressures.
Change from Baseline 24-hour Ambulatory Diastolic Blood Pressure at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  We will obtain continuous measures of diastolic blood pressure over a 24-h period with an FDA approved and European Society of Hypertension validated Non-Invasive Ambulatory Blood Pressure monitor. Blood pressure data will be broken into daytime (16 hour) and nighttime (8 hour) segments according to participants' individual sleep-wake cycles. Mean systolic and diastolic blood pressures (mmHg) will be calculated for the daytime and nighttime periods to evaluate circadian systolic and diastolic blood pressure profiles.
Change from Baseline Six-Minute Walk Distance at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  A six-minute walk test will be performed in a 30-meter hallway with cones to mark the ends of the track. The subject will be instructed to walk as quickly as they can, without running, for six minutes. They will start at the first cone and walk down the hallway, rounding the second cone, and returning up the hallway toward the first cone. They will continue to walk up and down the hallway, completing as many laps as possible in six minutes. Subjects will be told how much time is remaining every minute of the test, and with 30 seconds and 10 seconds remaining, and encouraged to walk as quickly as possible each time. Distance covered in six minutes will be recorded.
Change from Baseline NIH Toolbox - Cognitive Domain at 23 weeks, and 36 weeks | Measured at Baseline, Week 23, Week 36 to establish the intermediate and long-lasting effects of IMST
  Subjects will complete the 7 cognitive domain assessments from the NIH Toolbox for the Assessment of Neurological and Behavioral Function. These tests include: 1) flanker inhibitory control and attention test; 2) dimensional change card sort test; 3) list sorting working memory test; 4) picture sequence memory test; 5) oral reading recognition test; 6) picture vocabulary test; and 7) pattern comparison processing speed test. All tests will be performed on an iPad with an investigator presenting task instructions and monitoring compliance, as recommended by the American Academy of Neurology.
Change from Baseline Maximal Inspiratory Pressure at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  Maximal inspiratory pressure (PImax) will be assessed by having subjects generate 3 maximal inspiratory efforts against 3 cmH2O resistance measured at the mouth with a POWERbreathe™ KH2 trainer. If there is > 10% difference between efforts, subjects will perform up to 3 more efforts to ensure PImax is achieved. The average of the 3 greatest pressures.
Change from Baseline Resting Heart Rate at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  Resting heart rate will be measured simultaneously with blood pressure using the same automated oscillometric sphygmomanometer as is used for blood pressure assessments. As with blood pressure, heart rate will be defined as the average of the three readings.
Change from Baseline Home Sleep Apnea Testing at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  Severity of obstructive sleep apnea (i.e., AHI) will be assessed with a Nox T3s Home Sleep Apnea Testing diagnostic device, a Type III polygraph with actigraphy. Subjects will be instructed on the use and fitting of the device. They will be instructed to turn on the device immediately prior to going to bed and to turn it off upon waking. Subjects with an AHI < 15 will be excluded from the study. Outcomes include total sleep time, apneas/hour, hypopneas/hour, average O2 saturation (SpO2), minimum SpO2, duration of SpO2 < 90%, and duration of SpO2 < 85%.
Change from Baseline Grip Strength at 24 weeks, 28 weeks, and 36 weeks | Measured at Baseline, Week 24, Week 28, and Week 36 to establish the intermediate and long-lasting effects of IMST
  Maximal grip strength will be obtained with a Jamar hydraulic grip strength dynamometer. Handle position of the dynamometer will be standardized at position II. The subject will be seated with the shoulder in neutral position and the elbow supported and flexed to 90◦ with the forearm and wrist in neutral position. The subject will squeeze the dynamometer handle as hard as possible for 3 seconds and maximal force will be recorded in kg. The subject will perform three trials with each hand, and 15 seconds rest will be allowed between trials. Peak force of each hand will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth F Bailey, PhD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Respiratory and Neurophysiology Laboratory, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] DeLucia CM, DeBonis DR, Schwyhart SM, Bailey EF. Acute cardiovascular responses to a single bout of high intensity inspiratory muscle strength training in healthy young adults. J Appl Physiol (1985). 2021 Apr 1;130(4):1114-1121. doi: 10.1152/japplphysiol.01015.2020. Epub 2021 Feb 18. PMID 33600284
- [Background] Ramos-Barrera GE, DeLucia CM, Bailey EF. Inspiratory muscle strength training lowers blood pressure and sympathetic activity in older adults with OSA: a randomized controlled pilot trial. J Appl Physiol (1985). 2020 Sep 1;129(3):449-458. doi: 10.1152/japplphysiol.00024.2020. Epub 2020 Jul 30. PMID 32730174
- [Background] DeLucia CM, De Asis RM, Bailey EF. Daily inspiratory muscle training lowers blood pressure and vascular resistance in healthy men and women. Exp Physiol. 2018 Feb 1;103(2):201-211. doi: 10.1113/EP086641. Epub 2018 Jan 15. PMID 29178489
- [Background] Vranish JR, Bailey EF. Inspiratory Muscle Training Improves Sleep and Mitigates Cardiovascular Dysfunction in Obstructive Sleep Apnea. Sleep. 2016 Jun 1;39(6):1179-85. doi: 10.5665/sleep.5826. PMID 27091540
- [Background] Vranish JR, Bailey EF. Daily respiratory training with large intrathoracic pressures, but not large lung volumes, lowers blood pressure in normotensive adults. Respir Physiol Neurobiol. 2015 Sep 15;216:63-9. doi: 10.1016/j.resp.2015.06.002. Epub 2015 Jun 22. PMID 26112283
- [Derived] Tavoian D, Ramos-Barrera LE, Craighead DH, Seals DR, Bedrick EJ, Alpert JS, Mashaqi S, Bailey EF. Six Months of Inspiratory Muscle Training to Lower Blood Pressure and Improve Endothelial Function in Middle-Aged and Older Adults With Above-Normal Blood Pressure and Obstructive Sleep Apnea: Protocol for the CHART Clinical Trial. Front Cardiovasc Med. 2021 Nov 24;8:760203. doi: 10.3389/fcvm.2021.760203. eCollection 2021. PMID 34901220
- See also: Pre-screening questionnaire for interested participants — https://redcap.link/breathe